CLINICAL TRIAL: NCT07237399
Title: Percutaneous Thermo-ablation for the Treatment of Prostate Cancer Oligometastatasis (TA-P-OLIM): a Single Arm Phase II Study
Brief Title: Percutaneous Thermo-ablation for the Treatment of Prostate Cancer Oligometastatasis (TA-P-OLIM)
Acronym: TA-P-OLIM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0064
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Oligometastatic Prostate Cancer (OMPC); Prostate Cancer (Adenocarcinoma); Ablation Techniques
Keywords: thermal ablation; prostate cancer; cryoablation
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Transurethral Resection of Prostate; Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oligometastatic prostate cancer: The TA-P-OLIM Phase II study is a prospective, single-arm clinical trial designed to assess the safety, efficacy, and feasibility of percutaneous thermal ablation in the treatment of oligometastatic prostate cancer in patients who are no longer eligible for or refuse stereotactic body radiation therapy SBRT.
  Interventions: Procedure: Thermal ablation

INTERVENTIONS:
Procedure: Thermal ablation — Percutaneous thermal ablation is a minimally invasive technique that locally destroys tumor tissue using either heat (via microwave or radiofrequency ablation) or cold (via RFA ablation). Cryoablation is the most commonly used modality for this indication. It is generally well tolerated and enables precise treatment, as the ice ball created during the procedure can be continuously monitored using imaging, ensuring accurate tumor coverage while preserving surrounding healthy tissue.
  Other Names: cryoablation; RFA; MWA; radiofrequency ablation; microwave ablation; percutaneous thermal ablation

SUMMARY:
The TA-P-OLIM Study (Percutaneous Thermo-Ablation of Prostate Cancer OligoMetastasis) is a prospective, interventional phase II study designed to evaluate the feasibility, efficacy, and safety of percutaneous thermal ablation (TA) as a metastasis-directed therapy (MDT) for patients with oligometastatic prostate cancer. So far, these metastases have been locally treated with stereotactic body radiation therapy (SBRT) or surgical resection.

Percutaneous TA is a minimally invasive technique that locally destroys tumor tissue using either heat (via microwave or radiofrequency ablation) or cold (via cryoablation). This is achieved by inserting specialized needles into the tumor through a small skin incision under image guidance.

TA offers a valuable treatment option for patients who are not suitable candidates for SBRT, such as those with prior radiation exposure or metastases located near critical anatomical structures. In many of these cases, ablation remains feasible through the use of adjunctive thermoprotection techniques, where fluid is injected via a needle to gently displace critical structures, thereby creating a safe buffer zone during treatment.

Preliminary retrospective evidence shows that TA achieves comparable local tumor control rates to SBRT/resection with minimal complications.7 As a minimally invasive procedure, TA typically requires only a brief hospital stay-often on an outpatient basis-and enables rapid recovery. This makes TA an attractive alternative to surgery, which is associated with greater morbidity, longer recovery times, and limited suitability for some patients. In contrast to SBRT, TA also allows for simultaneous tissue sampling which is completed in a single session. Moreover, it can be safely repeated in the event of local recurrence.

The study focuses on patient-centered endpoints such as local control and tolerability, aiming to improve quality of life through personalized, minimally invasive treatment strategies. TA also offers an effective local treatment option for patients who are not eligible for standard treatments such as SBRT. In this way, an alternative to both SBRT and surgery is provided, enabling continued local treatment for patients.

Patients are eligible if they have previously received radical treatment for prostate cancer (surgery or radiotherapy, with or without hormonal therapy), subsequently developed a limited number of metastases (1-5), and are no longer candidates for or deny SBRT.

UZ Ghent, with its long-standing research expertise in metastasis-directed therapies for oligometastatic prostate cancer, coordinates the study. The project was established in collaboration with various departments within the Urological Multidisciplinary Tumor Board. Several centers in East and West Flanders have already confirmed their willingness to participate in the study.

ELIGIBILITY:
Inclusion criteria:

* > 18 years old
* PCa, treated with curative intent (radical prostatectomy, primary radiotherapy, or a combination of both) and oligorecurrent/oligopersistent metastasis (1 - 5 lesions) on imaging (PSMA-PET, CT, MRI).
* Recurrence or progression of metastases on imaging (PSMA-PET, CT, MRI) that cannot be treated with SBRT, either due to a history of previous high-dose radiotherapy with dose constraints, because SBRT is technically unfeasible or unsafe for the specific lesions, or because the patient refuses to undergo SBRT.
* PSMA-positive lesion
* Lesions up to 4 cm that are suitable and safe for TA with an anticipated high rate of technical success
* 'Eastern Cooperative Oncology Group' (ECOG) performance status of 2 or less.
* Patients can be androgen sensitive (mHSPC) or castration resistant (mCRPC).
* All patients will be discussed at the Multidisciplinary Tumor Board.

Exclusion criteria:

* <18y
* Severe comorbidity which limits the further life expectancy of the patient to < 2 years (opinion of the physician) and no malignancies < 2 years ago except for non-melanoma skin cancer and non-muscle invasive bladder cancer.
* No local radical treatment of the primary tumor was performed.
* Lack of compliance
* Absence of consent of the patient
* Location: intracranial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oligometastatic prostate cancer, characterized by 1-5 metastases who are no longer eligible for or refuse SBRT
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2031-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate | Until two years post treatment (thermal ablation)
  Proportion of patients without local progression of all treated lesions (multiple ablation sessions allowed) at 2 years, verified through follow-up imaging (PSMA-PET CT/CT/MRI) in at least 80% of patients.

SECONDARY OUTCOMES:
Tolerability of the treatment: proportion of patients without grade ≥3 treatment-related adverse events and without grade 5 adverse events following percutaneous ablative therapy | until 90 days post treatment
  This key secondary endpoint assesses treatment tolerability, defined as the proportion of patients without grade ≥3 treatment related adverse events and no grade 5 adverse events related to percutaneous ablative therapy at 30 and 90 days (according to Common Terminology Criteria for Adverse Events standards version 6)
Technical efficacy (feasibility) | 6 weeks post treatment
  Proportion of patients achieving complete ablation of all treated lesions on imaging 6 weeks post treatment.
Prostate-Specific Antigen progression-free survival (PSA-PFS) | Until 2 years post treatment
  Time from ablation to biochemical progression using PCWG3 criteria, that is,
  * if PSA ≥ 2 ng/mL at baseline: increase of ≥ 25% and ≥ 2 ng/mL.
  * if PSA < 2 ng/mL at baseline: increase of ≥ 25%.
PSA50 response | Until 2 years post treatment
  Proportion of patients achieving 50% decline in PSA from baseline at any time post-ablation.
Time to next-line systemic treatment-free survival (NEST-FS) | Until 2 years post treatment
  Time from ablation to initiation of new systemic treatment (androgen signaling inhibitor, chemotherapy, or other systemic therapy).
Distant progression-free survival (D-PFS) | Until 2 years post treatlent
  Time from ablation to identification of new distant metastasis on PSMA-PET/CT imaging.
Progression-free survival (PFS) | Until 2 years post treatment
  Time from ablation to first of the following: PSA progression, local or distant progression on imaging, start of new systemic therapy, death from any cause
Overall survival (OS) | Until two years post treatment
  Time from ablation to death from any cause.
Quality of Life assessed by the EORTC Quality of Life Questionnaire - Core 30 (QLQ-C30) | Until two years post treatment
  Quality of Life will be measured using the EORTC Quality of Life Questionnaire - Core 30 (QLQ-C30), a validated 30-item tool yielding scores from 0 to 100. For functioning scales and global health/QoL, higher scores indicate better functioning. For symptom scales and single-item symptom measures, higher scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No